CLINICAL TRIAL: NCT01005199
Title: Sorafenib Alone or in Combination With Everolimus in Patients With Unresectable Hepatocellular Carcinoma. A Randomized Multicenter Phase II Trial.
Brief Title: Sorafenib Tosylate With or Without Everolimus in Treating Patients With Localized, Unresectable, or Metastatic Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 77/08 and SASL 29; SWS-SAKK-77/08 (Other: SAKK); SWS-SASL-29; 2009-011884-35 (EudraCT Number); EU-20983; CDR0000657702
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Everolimus; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Sorafenib standard (Experimental): • Arm A (standard treatment): Sorafenib 2 x 400 mg daily until progressive disease, unacceptable toxicity, or consent withdrawal. (46 patients).
  Interventions: Drug: sorafenib tosylate
- Arm B: Sorafenib + everolimus (Experimental): • Arm B (investigational treatment): Sorafenib 2 x 400 mg daily plus everolimus 1 x 5 mg daily until progressive disease, unacceptable toxicity, or consent withdrawal. (60 patients)
  Interventions: Drug: everolimus; Drug: sorafenib tosylate

INTERVENTIONS:
Drug: everolimus — Sorafenib 2 x 400 mg daily plus everolimus 1 x 5 mg daily
  Other Names: RAD001
  Arms: Arm B: Sorafenib + everolimus
Drug: sorafenib tosylate — Sorafenib 2 x 400 mg daily
  Other Names: BAY 43-9006

SUMMARY:
RATIONALE: Sorafenib tosylate and everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This randomized phase II trial is studying giving sorafenib tosylate together with everolimus to see how well it works compared with sorafenib tosylate alone in treating patients with localized, unresectable, or metastatic liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if sorafenib tosylate with versus without everolimus can stop tumor progression in patients with localized, unresectable, or metastatic hepatocellular carcinoma.
* To evaluate changes in symptom-related and global quality of life (QL) and QL benefit over the course of trial treatment in these patients.
* To compare the primary endpoint (i.e., progression-free survival at week 12) to the QL benefit within 12 weeks from baseline.
* To evaluate how symptom-related and global QL indicators map on the single summary index derived from a standardized measure of health status for utility cost analysis.

OUTLINE: This is a multicenter study. Patients are stratified according to WHO performance status (0 vs 1), disease spread (extrahepatic spread vs non-extrahepatic spread), and center. Patients are randomized to 1 of 2 treatment arms.

* Arm A (standard treatment): Patients receive oral sorafenib tosylate twice daily for 4 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
* Arm B (investigational treatment): Patients receive oral sorafenib tosylate twice daily and oral everolimus once daily for 4 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Some patients may undergo CT scan or MRI at baseline and at 6 and 12 weeks during study to assess tumor response, tumor size, and tumor density.

Patients complete quality of life questionnaires at baseline and every 2 weeks for 12 weeks during study treatment.

After completion of study treatment, patients are followed every 2 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically, cytologically, or radiologically confirmed hepatocellular carcinoma (HCC)

  * Localized, unresectable, or metastatic disease
  * Child-Pugh class A or mildly decompensated Child-Pugh class B liver dysfunction (Child-Pugh score ≤ 7)
  * Stage B or C disease according to the Barcelona Clinic Liver Cancer (BCLC) staging classification
* Measurable disease

  * At least 1 unidimensionally measurable site of disease (≥ 10 mm in case of a non-nodal lesion or with a short axis ≥ 15 mm in case of a lymph node) by spiral/multi-slice CT/MRI scan according to revised RECIST criteria
* No locally advanced disease AND a candidate for radical surgery
* No known fibrolamellar HCC or mixed cholangiocarcinoma/HCC
* No clinical symptoms or history of CNS metastases or leptomeningeal disease (no imaging required)

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Hemoglobin ≥ 90 g/L
* Neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 75 x 10^9/L
* Creatinine clearance ≥ 40 mL/min
* ALT ≤ 5 times upper limit of normal
* INR ≤ 2
* Urine dipstick for proteinuria ≤ 1+ OR protein spot urine < 0.6 g/L
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study therapy
* No prior malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or localized nonmelanoma skin cancer
* No history of hemorrhagic or thrombotic cerebrovascular event within the past 12 months
* No documented variceal hemorrhage within the past 3 months
* No requirement for anticoagulant therapy except for low-dose anticoagulants for maintenance of patency of central venous access or prevention of deep vein thrombosis
* No history or presence of clinically significant acute or unstable cardiovascular, cerebrovascular, renal, gastrointestinal, pulmonary, endocrine, central nervous system, or immunological disorders (except for the presence of hepatitis B or C virus or cirrhosis) within the past 6 months
* No encephalopathy
* No known HIV infection
* No active infection requiring IV antibiotics
* No arterial hypertension ≥ 150/100 mm Hg despite therapy
* No ongoing cardiac dysrhythmias of NCI CTCAE grade ≥ 2, atrial fibrillation of any grade, prolongation of QTc > 500 msec on screening electrocardiogram (ECG), or history of familial long QT syndrome
* No repeated paracentesis (more than 1 per month)
* No psychiatric disorder precluding understanding of information of trial-related topics, giving informed consent, or interfering with compliance for oral drug intake
* No concurrent grapefruit, grapefruit juice, or products containing bitter oranges
* Able to take oral medications
* Completed baseline quality of life questionnaire
* Must be compliant and geographically proximal for follow-up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic anticancer treatment for this disease

  * The following prior therapies are allowed provided previously treated lesions remain separate from those to be measured in the current trial and prior treatment is completed within the past 4 weeks

    * Surgery
    * Liver-directed therapy (e.g., transarterial embolization/chemoembolization [limited to 5 treatments], radiofrequency ablation, cryoablation, radiotherapy, or percutaneous ethanol injection)
* No prior organ transplantation
* No concurrent estrogen-containing supplementary therapy
* No concurrent full-dose anticoagulation with coumarin derivatives
* No concurrent elective major surgery
* No concurrent radiotherapy (concurrent analgesic radiotherapy of non-target lesions allowed)
* No concurrent or anticipated need for CYP3A4 inhibitors or inducers, unless the drugs are medically necessary and no substitutes are available, including any of the following:

  * Ketoconazole
  * Itraconazole
  * Voriconazole
  * Erythromycin
  * Clarithromycin
  * Diltiazem
  * Verapamil
  * Protease inhibitors
* No concurrent strong CYP3A4 inducers*, including any of the following:

  * Carbamazepine
  * Continuous dexamethasone (> 2 mg/day for > 7 days)
  * Phenobarbital
  * Phenytoin
  * Rifampicin
  * St. John's wort NOTE: *Concurrent antacids allowed provided they are administered > 1 hour before or > 1 hour after trial drug administration.
* No other concurrent experimental drugs or anticancer therapy or treatment in another clinical trial within the past 30 days
* No other concurrent investigational drugs
* No chronic systemic steroids or other immunosuppressive agents
* No concurrent angiotension converting enzyme inhibitors (ACE-I)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2009-11; Primary Completion 2013-06 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | at 12 weeks

SECONDARY OUTCOMES:
Objective response | during trial treatment and follow-up (max. 3 years)
Disease stabilization (DS) | under trial treatment
Duration of disease stabilization | Duration of DS (CR, PR or SD) will be calculated from the time that measurement criteria are met for the first time until documented tumor progression.
Progression-free survival (PFS) | PFS will be calculated from randomization until documented tumor progression or death, whichever occurs first
Time to progression (TTP) | TTP will be calculated from randomization until documented tumor progression or tumor-related death
Overall survival | from randomization until death
Adverse events at baseline and during trial treatment | All AEs will be assessed according to NCI CTCAE v3.0.
Serum alpha fetoprotein (AFP) level | Serum AFP levels will be measured during the therapy, if AFP is ≥ 1.5 x ULN at baseline.
Viral reactivation in patients with chronic hepatitis B or C virus infection | Number of patients with HCV/HBV (re)-activation during trial treatment
Correlation between vitamin B12 and overall survival | The baseline vitamin B12 value, collected at trial randomization, is correlated to overall survival when dichotomized by the cut-point of 600 ng/L.

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Koeberle, MD, Study Chair — Cantonal Hospital of St. Gallen; Jean-Francois Dufour, MD, Study Chair — Insel Gruppe AG, University Hospital Bern; Gyorgy Bodoky, MD, PhD, Study Chair — Szent Laszlo Korhaz; Michael Montemurro, MD, Study Chair — CHUV Lausanne
Locations (15):
- Medizinische Universität Wien, Vienna, Austria
- Szent Laszlo Korhaz, Budapest, Hungary
- Switzerland (13):
  - Saint Claraspital AG, Basel
  - Clinical Cancer Research Center at University Hospital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Bruderholz, Bruderholz
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Liestal, Liestal
  - Kantonsspital - St. Gallen, Sankt Gallen
  - CHCVS - Hôpital de Sion, Sion
  - Regionalspital, Thun
  - City Hospital Triemli, Zurich
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koeberle D, Dufour JF, Demeter G, Li Q, Ribi K, Samaras P, Saletti P, Roth AD, Horber D, Buehlmann M, Wagner AD, Montemurro M, Lakatos G, Feilchenfeldt J, Peck-Radosavljevic M, Rauch D, Tschanz B, Bodoky G; Swiss Group for Clinical Cancer Research (SAKK). Sorafenib with or without everolimus in patients with advanced hepatocellular carcinoma (HCC): a randomized multicenter, multinational phase II trial (SAKK 77/08 and SASL 29). Ann Oncol. 2016 May;27(5):856-61. doi: 10.1093/annonc/mdw054. Epub 2016 Feb 15. PMID 26884590